CLINICAL TRIAL: NCT01165801
Title: Size Progression of Non-Exudative Age-Related Macular Degeneration After Cataract Surgery
Brief Title: Size Progression of Macular Degeneration After Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EKAM-1-2061
Record Dates: First submitted 2010-07-17; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Cataract surgery; Size of AMD; Influence of cataract surgery on AMD Size
MeSH Terms: conditions — Macular Degeneration | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control Group (CO) (No Intervention): Fifty-four patients with cataract and non-exudative age-related macular degeneration (AMD) were randomized into an early surgery group (ES=28) with immediate cataract surgery and a control group (CO=26) where surgery was performed after six months.
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery — Fifty-four patients with cataract and non-exudative age-related macular degeneration (AMD) were randomized into an early surgery group (ES=28) with immediate cataract surgery and a control group (CO=26) where surgery was performed after six months.

SUMMARY:
The purpose of this study was to find out if in patients with non-exudative age-related macular degeneration (AMD), randomly assigned to cataract surgery, any AMD size progression or progression to exudative AMD could be detected 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and non-exudative age-related macular degeneration

Exclusion Criteria:

* Patients with retinal pathologies other than AMD, exudative AMD, progressive glaucoma, myopia > 10 diopters, panretinal laser treatment, former cataract or vitreoretinal surgery, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2002-01; Primary Completion 2007-09 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
AMD size (defined central region of interest) | at enrollment, after 6 months
  To evaluate AMD size progression, absolute and relative differences in pixels of the ROI were cal-culated by equivalent tests.

SECONDARY OUTCOMES:
Functional ophthalmic assessments | at enrollment, after 6 months
  Cataract grade (LOCS-III), Visual acuity (distance/near), contrast acuity tests, Visual Function Index (VF-14)

CONTACTS AND LOCATIONS:
Locations (1):
- The Rudolph Foundation Hospital, Dept. of Ophthalmology, Vienna, Vienna, Austria